CLINICAL TRIAL: NCT06419023
Title: Influence of Pilates Method Intervention on Changes in Myofascial Stiffness, Cardiorespiratory Fitness and Quality of Life in Women With Breast Cancer
Brief Title: Impact of Pilates Method on Myofascial Stiffness, Cardiorespiratory Fitness and Quality of Life in Breast Cancer Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MTarnas_PhD
Record Dates: First submitted 2024-05-06; First posted 2024-05-17 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Female
Keywords: Pilates Method; quality of life; myofascial stiffness; pain; cardiorespiratory fitness; inflammation; breast cancer; aromatase inhibitor
MeSH Terms: conditions — Pain; Inflammation; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises group (EG) (Experimental): The exercise group (EG) participated in supervised physical activity intervention using the Pilates Method (exercises on the mat, 60min each session, 2 sessions each week over 12 weeks) were administered by certified Pilates teacher.
  Interventions: Behavioral: supervised physical activity intervention using the Pilates Method (exercises on the mat)
- Usual-Care Group (U-CG) (No Intervention): Patients in the U-CG were instructed to continue with their usual activities: a) to avoid changing their diet habits during intervention; b) being physically active as usual.

INTERVENTIONS:
Behavioral: supervised physical activity intervention using the Pilates Method (exercises on the mat) — Each Pilates session was consisted of: a) introduction to the goal of training, familiarizing new skills (2-3 min); b) Pre-Pilates warm-up and respiratory exercises (5-10 min); c) mat Pilates exercises with the traditional Pilates repertoire: basic, beginner (40 min); d) cool down and endings exercises (5 min); e) session summary (2-3min). When required, exercises were adapted for breast cancer body needs and restrictions. Depending on the purpose of the exercise, different equipment was used (Pilates small ball 22 cm, Swiss ball, small massage balls, resistance band, towels, rollers, boxes, "Magic Circle").
  Arms: Exercises group (EG)

SUMMARY:
The effectiveness of breast cancer treatment is quite well documented. Still, side effects can underpin other treatment-induced diseases such as osteopenia, diabetes, and especially cardiovascular dysfunction. Therefore, finding a method that could partly counteract these side effects and at the same time be implemented throughout treatment is a challenge for researchers.

The main purpose of this experimental, randomized control trial was to analyze the effect of the Pilates Method (PM) intervention on changing the myofascial stiffness along the thoracic and lumbar spine, cardiorespiratory fitness and quality of life in women with breast cancer receiving aromatase inhibitor therapy. The apllied procedure of 12 -week PM training included the training intervention based on hypothesis:

* PM reduces myofascial stiffness along the thoracic and lumbar spine of women with breast cancer receiving aromatase inhibitor therapy
* PM improves the cardiorespiratory fitness of women with breast cancer receiving aromatase inhibitor therapy
* PM improves the quality of life of women with breast cancer receiving aromatase inhibitor therapy.

Possible practical applications include the domains of exercise medicine, physical activity in cancer and public health.

DETAILED DESCRIPTION:
The trial was conducted by Poznan University of Physical Education in cooperation with UMP (Poland).

This design of trial assumed the parallel two-arm group, prospective, randomized controlled trial (RCT) comparing an exercises-based intervention (experimental group) to usual care and physical activity recommendation (control group) in women with breast cancer with perioperative hormonal treatment AI.Randomization were performed as a simple randomization with a 1:1 allocation (coin toss).

All patients were assessed and recruited by two oncologists regarding eligibility to participate in the study.

Before enrollment, all participants were given detailed information about experiment, procedures, risks, and benefits of the study and gave their written consent to participation. The patients were informed at any stage of the project may resign from participation without having to give a reason.The study was conducted in two stages. Patient recruitment and data collection started in February 2022. The baseline assessment of patients is carried out two weeks before the start of PT intervention. PT intervention lasted 12 weeks. Post-intervention assessment is performed during two weeks after PT intervention. Finally data (reports) collection and data preparation for analysis were completed in December 2023.

Potential patients matching primary criteria underwent clinical, laboratory, EKG and echocardiographic follow-up assessment by cardiologist. Clinical specialists eligible for the study provided information about the study and presented informed consent to patients. The patients were referred for further study diagnostics after clinical qualification and signed written informed consent to the planned research.

Together with oncologists the research group also included sports physiologists, cardiologist, certified Pilates teacher. All participants were evaluated by same qualified personnel according to standardized test protocols and in the same conditions at baseline and after 12-week intervention. Objective physical measurements were performed by trained and blinded assessors unaware of the assignment information.

At the baseline and post training period were performed following assessments:

* anthropometrics using digital stadiometer
* body composition tested by the dual X-ray absorptiometry method
* bone mineral density tested by the dual X-ray absorptiometry method
* questionnaire assessment of: (i) quality of life using EORTC QLQ-C30 Questionnaire version 3.0, EORTC QLQ-BR23 Questionnaire Breast cancer module), (ii) pain using Brief Pain Inventory Short Form Questionnaire), (iii) level of physical activity using IPAQ Questionnaire
* myofascial stiffness using myotonometr and a non-invasive shear-wave elastography examination
* respiratory function measured with spirometric tests
* cardiorespiratory fitness measured with: (i) cardiopulmonary exercise test CPET on the treadmil, (ii) metabolic response assessment with blood lactic acid concentration, (iii) subjective rating of perceived exertion with the Borg 6-20 scale
* vascular circulation indicators measured with the use of the Flow Mediated Skin Fluorescence
* inflammatory hematological ratios were calculated based on hematological medical patients indicators.

Patients characteristics has been completed by medical records and socio-demographic questionnaires.

The supervised physical activity intervention using the Pilates Method (60min each session, 2 sessions each week over 12 weeks) was used in this study.

In the study took part two groups - Exercise Group (experimental group performing PM intervention) and Usual-Care Group (control group).

The training program involved exercise performed on mats. The subjects took part in a model training session, during which all exercises were explained, performance was discussed, common mistakes were pointed out, and efforts were made to maintain proper exercise intensity and muscle activation and relaxation.The model PM training sessions was consisted of:

1. warm-up and respiratory exercises (5-10 min);
2. mat Pilates exercises with the traditional Pilates repertoire (basic, beginner) adapted for breast cancer patients needs and restrictions (40 min);
3. cool down and endings exercises (5 min);
4. session summary (2-3min). The training program was supervised by the same specialist of PM.

ELIGIBILITY:
Inclusion Criteria:

1. women with invasive breast cancer
2. stage of disease according to TNM classification I-III
3. cancer with estrogen receptor expression in at least 10% of cell nuclei
4. supplemental hormone therapy with an aromatase inhibitor used for at least 6 months
5. performance status according to ECOG classification 0-1
6. BMI of 18.5-30
7. without chronic diseases affecting the limitation of the use of oncological treatment
8. without contraindications to participation in group supervised Pilates classes
9. participation in at least 17 of 24 classes according to the proposed schedule

Exclusion Criteria:

1. invasive breast cancer stage IV according to TNM classification
2. performance status according to ECOG classification 2-4
3. unregulated hypertension
4. unstable ischemic heart disease
5. arrhythmia
6. rheumatic diseases
7. osteoporosis
8. advanced osteoarthritis
9. disease of rheumatic origin (AS, RA, fibromyalgia)
10. pregnancy
11. BMI < 18.5 or above 30
12. unregulated hypothyroidism/hyperthyroidism

Criteria for drop out The criteria for discontinuing allocated interventions are as follows: 1) participant's voluntary withdrawal from the study; 2) worsening of oncological prognosis that prevents the continuation; 3) absence of training sessions due to unjustified reasons in the case of the PG (compliance below 70%).

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Quality of life - Global Health Status | before and after 12-week intervention
  Quality of life - Global Health Status (GHS) assessment with EORTC QLQ-C30 Questionnaire version 3.0. On the scale minimum value is 1, maximum value is 7. A high score represents a high QoL (better outcome).
Quality of life - Functional scores | before and after 12-week intervention
  Quality of life - Functional scores assessment with EORTC QLQ-C30 Questionnaire version 3.0.
  On the scale minimum value is 1, maximum value is 4. A high score represents a high /healthy level of functioning (better outcome).
Quality of life - Symptom scores | before and after 12-week intervention
  Quality of life - Functional scores assessment with EORTC QLQ-C30 Questionnaire version 3.0.
  On the scale minimum value is 1, maximum value is 4. A high score for a symptom scale represents a high level of symptomatology /problems (worse outcome).
Quality of life - Functional scores (body image, sexual functioning, sexual enjoyment, future perspective) | before and after 12-week intervention
  Quality of life - Functional scores (body image, sexual functioning, sexual enjoyment, future perspective) assessment with EORTC QLQ-BR23 Questionnaire (Breast cancer module). On the scale minimum value is 1, maximum value is 4. A high score represents a high /healthy level of functioning (better outcome).
Quality of life - Symptom scores (systemic therapy side effects, breast symptoms, arm symptoms, upset by hair loss) | before and after 12-week intervention
  Quality of life - Symptom scores (systemic therapy side effects, breast symptoms, arm symptoms, upset by hair loss) assessment with EORTC QLQ-BR23 Questionnaire (Breast cancer module).On the scale minimum value is 1, maximum value is 4. A high score for a symptom scale represents a high level of symptomatology / problems (worse outcome).
Subjective pain assessment - Pain Severity Total Score | before and after 12-week intervention
  Pain Severity Total Score assessment with Brief Pain Inventory (short form) Questionnaire. Pain severity is measured by four items: worst pain, least pain, average pain in the last 24 h, and pain now. On the scale minimum value is 0 (no pain), maximum value is 10 (pain as as you can imagine).
Subjective pain assessment - Pain Interference Total Score, Physical Interference, Affective Interference | before and after 12-week intervention
  Pain Interference Total Score, Physical Interference, Affective Interference assessment with Brief Pain Inventory (short form) Questionnaire. The seven interference items (sleep disturbance, general activity, mood, work, relations with others, walking, and enjoyment of life) are assessed on a 0 to 10 scale, with 0 being "did not interfere" and 10 being "interfered completely".
Subjective pain assessment - the extent of pain complaints | before and after 12-week intervention
  The extent of pain complaints assessment with Brief Pain Inventory (short form) Questionnaire. Pointing out on the body diagram the places where the subject feels pain.
Myofascial stiffness | before and after 12-week intervention, before and after unit Pilates session
  Myofascial stiffness (N/m) assessment using myotonometer, MyotonPro® .
Myofascial stiffness | before and after 12-week intervention
  Assessment of myofascial stiffness (kPa) and (m/s) using a non-invasive shear-wave elastography examination AIXPLORER SuperSonic Imagine.
Resting Vital Capacity | before and after 12-week intervention
  Level of Resting Vital Capacity (l). Respiratory function assessment using MetaMax 3B-R2, MetaSoft Studio software 5.1.0, Cortex Biophysics Gmhb, Leipzig, Germany.
Forced Vital Capacity | before and after 12-week intervention
  Level of Forced Vital Capacity (l). Respiratory function assessment using MetaMax 3B-R2, MetaSoft Studio software 5.1.0, Cortex Biophysics Gmhb, Leipzig, Germany.
Maximal Voluntary Ventilation | before and after 12-week intervention
  Maximal Voluntary Ventilation (l/min). Respiratory function assessment using MetaMax 3B-R2, MetaSoft Studio software 5.1.0, Cortex Biophysics Gmhb, Leipzig, Germany.
Forced Expiratory Volume in the first second of expiration | before and after 12-week intervention
  Forced Expiratory Volume in the first second of expiration in %. Respiratory function assessment using MetaMax 3B-R2, MetaSoft Studio software 5.1.0, Cortex Biophysics Gmhb, Leipzig, Germany.
Peak Expiratory Flow | before and after 12-week intervention
  Peak Expiratory Flow (l/s). Respiratory function assessment using MetaMax 3B-R2, MetaSoft Studio software 5.1.0, Cortex Biophysics Gmhb, Leipzig, Germany
The modified Tiffeneau-Pinelli index | before and after 12-week intervention
  The modified Tiffeneau-Pinelli index is Forced Expiratory Volume in 1 second/ Vital Capacity ratio (%). A ratio below 70% is typically indicative of obstructive lung disease. Respiratory function assessment using MetaMax 3B-R2, MetaSoft Studio software 5.1.0, Cortex Biophysics Gmhb, Leipzig, Germany.
absolute Oxygen Uptake | before and after 12-week intervention
  Absolute Oxygen Uptake (l/min) at rest, at anaerobic threshold (AT), at respiratory compensation point (RCP). Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
relative Oxygen Uptake | before and after 12-week intervention
  Relative Oxygen Uptake (l/min/kg) at rest, at anaerobic threshold (AT), at respiratory compensation point (RCP). Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Volume of carbon dioxide | before and after 12-week intervention
  Volume of carbon dioxide (l/min) at rest, at anaerobic threshold (AT), at respiratory compensation point (RCP). Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
absolute Power Output | before and after 12-week intervention
  Absolute Power Output (Watts) at rest, at anaerobic threshold (AT), at respiratory compensation point (RCP), at maximal/peak oxygen uptake. Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
relative Power Output | before and after 12-week intervention
  Relative Power Output (W/kg) at rest, at anaerobic threshold (AT), at respiratory compensation point (RCP), at maximal/peak oxygen uptake. Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Power Output when respiratory ratio (RQ) equal 1 | before and after 12-week intervention
  Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Ventilatory equivalent for carbon dioxide | before and after 12-week intervention
  Ventilatory equivalent for carbon dioxide (l/min) Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Minute ventilation per carbon dioxide production VE/VCO2 slope | before and after 12-week intervention
  Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Heart Rate | before and after 12-week intervention
  Resting and maximal Heart Rate (beats/min). Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while an walking test on the treadmill using a heart rate monitor.
Blood Lactic Acid Concentration | before and after 12-week intervention
  Metabolic response assessment with blood lactic acid concentration (mmol/l) are tasted before and after a cardiopulmonary exercise test (CPET) (Biosen C-line, EKF Diagnostics)
Subjective rating of perceived exertion | before and after 12-week intervention
  Borg 6-20 scale was applied to indicate the level of exertion by participant at maximal oxygen uptake /peak oxygen uptake workload during CPET. On the scale minimum value is 6 (no exertion at all), maximum value is 20 (maximal exertion).

SECONDARY OUTCOMES:
Body Height | before and after 12-week intervention
  Body Height (m) is measured using Digital stadiometer (Seca 285, SECA, Hamburg, Germany).
Body Mass | before and after 12-week intervention
  Body Mass (kg) is measured using Digital stadiometer (Seca 285, SECA, Hamburg, Germany).
Total Body Mass | before and after 12-week intervention, test conducted while fasting
  Total Body Mass (kg). Indicators of body composition are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Bone Mass | before and after 12-week intervention, test conducted while fasting
  Bone Mass (kg). Indicators of body composition are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Muscle Mass | before and after 12-week intervention, test conducted while fasting
  Muscle Mass (kg). Indicators of body composition are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Skeletal Muscle Mass | before and after 12-week intervention, test conducted while fasting
  Skeletal Muscle Mass (kg). Indicators of body composition are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Lean Body Mass | before and after 12-week intervention, test conducted while fasting
  Lean Body Mass (kg). Indicators of body composition are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Fat Mass | before and after 12-week intervention, test conducted while fasting
  Fat Mass (kg). Indicators of body composition are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Fat-Free Mass | before and after 12-week intervention, test conducted while fasting
  Fat-Free Mass (kg). Indicators of body composition are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Visceral Adipose Tissue 1 | before and after 12-week intervention, test conducted while fasting
  Visceral Adipose Tissue (cm^3). Indicators of body composition are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Visceral Adipose Tissue 2 | before and after 12-week intervention, test conducted while fasting
  Visceral Adipose Tissue (g). Indicators of body composition are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Body Mass Index | before and after 12-week intervention, test conducted while fasting
  Body Mass Index (BMI) (kg/m^2). Indicators of body composition are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Relative Skeletal Muscle Mass Index | before and after 12-week intervention, test conducted while fasting
  Relative Skeletal Muscle Mass Index (RSMI) (kg/m^2). Indicators of body composition are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Intra-Cellular Water | before and after 12-week intervention, test conducted while fasting
  Intra-Cellular Water (kg). Body water component measured using TANITA MC-98OMA plus device.
Extra-Cellular Water | before and after 12-week intervention, test conducted while fasting
  Extra-Cellular Water (kg). Body water component measured using TANITA MC-98OMA plus device.
Total Body Water | before and after 12-week intervention, test conducted while fasting
  Total Body Water (kg). Body water component measured using TANITA MC-98OMA plus device.using TANITA MC-98OMA plus device.
Bone Mineral Density | before and after 12-week intervention, test conducted while fasting
  Bone Mineral Density (g/cm^2). Indicators of bone mineral density are tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Bone Mass Component | before and after 12-week intervention, test conducted while fasting
  Bone Mass Component (kg). Indicator is tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
T-Score | before and after 12-week intervention, test conducted while fasting
  T-Score Index. Indicators of bone mineral density are tested and calculated by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Z-Score | before and after 12-week intervention, test conducted while fasting
  Z-Score Index. Indicators of bone mineral density are tested and calculated by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA and enCORE v. 16 SP1 software).
Inflammatory hematological ratios | before and after 12-week intervention
  Indicators of inflammation (Neutrophil to Lymphocyte ratio, Monocyte to Lymphocyte ratio, Platelet to Lymphocyte ratio) are calculated made based on hematological medical records.
Level of Physical activity | before and after 12-week intervention
  A self-report scale that measures physical activity. The IPAQ comprises 27 items that assess time spent engaging in various levels of physical activity and includes sitting time. Participants are asked to report their responses in terms of minutes, hours, or days. The units of measurement are METs min/week. The amount of physical activity is assessed based on intensity (moderate, intense, walking), and the amount of total physical activity is calculated by summing up the records across each dimension by intensity. A category of low physical activity is considered a result in the total physical activity below 600 METs min/week, moderate between 600 and 3000 METs min/week and high above 3000 METs min/week. Scores can be computed continuously or categorically.
Oxygen Pulse | before and after 12-week intervention
  Oxygen Pulse (ml). Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Breathing Frequency | before and after 12-week intervention
  Breathing Frequency (breaths/min). Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Respiratory Exchange Ratio | before and after 12-week intervention
  Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Ventilatory Efficiency | before and after 12-week intervention
  Ventilatory Efficiency (l/min) Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Tidal Volume | before and after 12-week intervention
  Tidal Volume (l) Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Speed | before and after 12-week intervention
  Speed (km/h). Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Distance | before and after 12-week intervention
  Distance (m) Indicators of aerobic capacity assessment with cardiopulmonary exercise test (CPET) is conducted while a test on the treadmill (H/P Cosmos Pulsar, Sports & Medical, Nussdorf-Traunstein, Germany) using a breath-by-breath ergospirometer (Metamax 3B R2ergospirometer and Metasoft Studio v. 5.1.0 software package Cortex Biophysik, Leipzig, Germany).
Indicators of vascular circulation | baseline (before and immediately after CPET) and after 12-week intervention (before and immediately after CPET)
  Vascular circulation indicators (Reactive Hyperemia Response, Hypoxia Sensitivity, Normoxia Oscillatory Index, the rate of Nicotinamide Adenine Dinucleotide fluorescence growth) are measured with the use of the Flow Mediated Skin Fluorescence (FMSF) using The AngioExpert device (AngioExpert, Poland).

OTHER OUTCOMES:
Clinical history | before and after 12-week intervention
  Patients clinical history are collected with study-specific questionnaires and medical records.
Socio-demographic characteristics | before 12-week intervention
  Socio-demographic characteristics are collected with study-specific questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Tarnas, Master, Principal Investigator — Department of Athletics, Strength and Conditioning, Poznan Univ of Physical Ed, Poland
Locations (1):
- Poznan University of Physical Education, Poznan, Greater Poland Voivodeship, Poland